CLINICAL TRIAL: NCT00743223
Title: The Frequency Forward Head Posture in Subjects With Temporomandibular Disorder
Status: Completed | Type: Observational
Sponsor: Federal University of Mato Grosso (Other)
Responsible Party: GUSTAVO HELDER VINHOLI, Federal University of Mato Grosso do Sul
Other Study IDs: CEP-UNIFESP1175/06
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2008-08-28 (Estimated); Status verified 2008-08

CONDITIONS: Temporomandibular Disorder
Keywords: temporomandibular disorder; orofacial pain; posture of the head
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Study-group: The volunteers were selected on a randomized form among the individuals who went to the clinic of orofacial pain and temporomandibular disorders of São Paulo Hospital.
  Interventions: Other: The measure of the cervical posture
- 2: Control-group: The volunteers were selected on a randomized form among the individuals who went to the dental offices of the researchers.
  Interventions: Other: The measure of the cervical posture

INTERVENTIONS:
Other: The measure of the cervical posture — The investigation of the cervical position consisted of locating the individual in side view with the parallel feet in erect position and tracing an imprisoned plumb wire to the ceiling and tangent to the kyphosis curve of the thoracic column. With a ruler it was verified at a distance of this line until the point deepest of the cervical lordosis curve.
  Other Names: there are not brand or serial numbers.

SUMMARY:
The aim of this study was to verify the frequency of the forward head posture in subjects with temporomandibular disorder and to compare them with control group

DETAILED DESCRIPTION:
Postural habit is defined as "the attitude of the body" being characterized as good when the parts of the body muscles and bones are lined up and work together in a harmonious form protecting the body of injury or gradual deformity and independently the attitude. The bad posture is a bad habit, but it can be which results in the disagreement of some parts of the body. These are at risk of injury or pain due to and increased tension that the disagreement imposes to the support structures. Several study confirm this occurrence relating that this the attitude can alter itself principally if a discomfort occurs. When it occurs there will be the installation of alterations, limitation of movements or even deformity, leading it to the development of an abnormal of posture of the body which will be able to reduce the functional capacity of various structures and organs of the human body.

The forward head posture is a common abnormality in cervical spine that can contribute to perpetuation the trigger points in muscles of the head as well as some kinds of temporomandibular disorder. It was suggested its influence in the treatment of patients with orofacial pain and TMD the FHP may occur a result of an acute trauma or if develop itself gradually because of an inadequate position.

ELIGIBILITY:
Inclusion Criteria:

Study group

The criteria of inclusion of the individuals for this group were:

* Individuals whose main complaint were pain in the muscles of the chew or the TMJ
* To present pain of the muscle or to articulate during the functional tests
* Maximum opening interincisal equal or minor than 40 mm

Crontrol group

The criteria of inclusion of the individuals for this group were:

* Individuals who underwent routine dental treatment
* Individuals without TMD complaint
* Maximum opening interincisal bigger than 40 mm

Exclusion Criteria:

* There are not

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was randomized with one hundred subjects that were divided fifty for study group and fifty of the control group with age between 18 and 65 years old, of both sexes. The volunteers were selected among the individuals who went to the clinic of orofacial pain and TMD of São Paulo Hospital and the dental offices of the researchers
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-10; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Outcome Measure: frequency of the forward head posture | one year

CONTACTS AND LOCATIONS:
Overall Officials: GUSTAVO VINHOLI, DENTIST, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Barros TP, Campolongo GD, Novaes AP, Amantéa DV. The importance of the postural evaluation in patients with temporomandibular joint dysfunction. Acta ortop. Bras, 2004;12(3),jul/set:155-59 — http://www.bireme.br